CLINICAL TRIAL: NCT03907995
Title: Peer-led Group Intervention for Coping With Disaster
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: American National Red Cross (Other)
Responsible Party: Principal Investigator, Eric Alan Storch, Professor, Baylor College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-44353
Record Dates: First submitted 2019-04-04; First posted 2019-04-09 (Actual); Last update posted 2020-05-27 (Actual); Status verified 2020-05

CONDITIONS: Anxiety Disorder; PTSD; Depressive Symptoms; Anger; Depressive Disorder
MeSH Terms: conditions — Anxiety Disorders; Stress Disorders, Post-Traumatic; Depression; Depressive Disorder | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cognitive Behavioral Therapy (Experimental): The form of treatment will involve 6 group sessions every two weeks about an hour each. Sessions consist of teaching a different coping technique in each session to help cope with disaster or other events.
  Interventions: Behavioral: Cognitive Behavioral Therapy

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy — The form of treatment will involve 6 group sessions every two weeks about an hour each. Sessions consist of teaching a different coping technique in each session to help cope with disaster or other events.
  Other Names: Skills for Psychological Recovery; CBT

SUMMARY:
The present project partners with leading faith communities in Houston to provide expert-led educational workshops to a diverse sample of adults on normative and concerning response to disaster. Secondly implementing peer-led interventions where a trained adult leads others through an evidence-based manualized intervention. Lastly, identifying and referring individuals who require more intensive services to a higher level of care.

DETAILED DESCRIPTION:
Approximately 20% of individuals have significant behavioral health concerns. Exposure to a disaster like Hurricane Harvey and its aftermath often exacerbates pre-existing issues and/or brings new issues, with post-traumatic stress presenting in manners such as anxiety, depression, conduct issues and/or somatic issues. Approaches are needed that educate community members about both normative and concerning responses to disaster focused on coping skills development. A particular approach, peer-led intervention groups have been shown effective at delivering these types of intervention. Brief, psycho-educational peer-led programs have shown effectiveness in a variety of forums including helping promote adjustment among those who have experienced trauma. There will be six group sessions every two weeks. Sessions will include how to teach appropriate coping techniques to respond to the distress, confronting distressing memories related to the disaster, and emotion regulation techniques. After the group sessions end, individuals who require a more intensive service will be referred to a higher level of care.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older and English speaking.

Exclusion Criteria:

* Individuals under the age of 18 and non-English speaking and participants who do not wish to participate in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2019-05-29 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
PTSD Symptom Scale - Adult | Post-treatment, which is 12 weeks after baseline.
  The PTSD Symptom Scale - Self Report is a 17-item, Likert-scale, self-report questionnaire designed to assess the symptoms of PTSD according to DSM-IV. Each of the 17 items is rated on a scale from 0 to 3, with total score ranging from 0 to 51 by adding them up.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Storch, Ph.D., Principal Investigator — Baylor College of Medicine
Locations (1):
- Baylor College of Medicine: Jamail Specialty Care Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No